CLINICAL TRIAL: NCT06521645
Title: The Effect of Acupoint Stimulation on Level of Lactate in Patients Undergoing Cerebral Endovascular Intervention
Brief Title: Effect of Acupoint Stimulation on Lactate During Cerebral Endovascular Intervention
Acronym: ASLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJH-A-20240626
Record Dates: First submitted 2024-07-04; First posted 2024-07-26 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Endovascular Procedures
Keywords: acupoint stimulation; cerebral endovascular intervention; lactate
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupoint stimulation (Experimental): needles are inserted into the skin of Baihui acupoint, and electrical acupoint stimulation is given
  Interventions: Other: electroacupuncture
- Control (Sham Comparator): needles are shallowly inserted into the skin of Bihui acupoint, but no electrical acupoint stimulation is given
  Interventions: Other: sham needle

INTERVENTIONS:
Other: electroacupuncture — electrical stimulation is given through needles inserted into the skin
  Arms: Acupoint stimulation
Other: sham needle — needles are inserted shallowly into the skin
  Arms: Control

SUMMARY:
It is advocated that neuroprotection should be increased before endovascular treatment and that the penumbra should be protected from reperfusion damage after recanalization. Monitoring lactate and pH levels in acute ischemic stroke patients who have had endovascular recanalization can be utilized to predict mortality and morbidity, especially in the first five hours after the procedure. This study aims to observe the effect of acupoint stimulation on lactate level during endovascular recanalization.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* scheduled for cerebral endovascular intervention

Exclusion Criteria:

* American Society of Anesthesiologists status over level three
* history of cerebral vascular intervention
* history of severe neurological disease (stroke, neurological degenerative disease, psychiatric disease)
* severe hepatic or renal dysfunction
* severe glucose disorder or thyroid dysfunction
* contraindications to transcutaneous electrical stimulation (infection or injury of the skin area, implanted electrical devices)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
arterial level of lactate at 30 minutes after recanalization | 30 minutes after recanalization

SECONDARY OUTCOMES:
arterial level of lactate immediately after recanalization | about 1 minute after recanalization
pH value at 30 minutes after recanalization | 30 minutes after recanalization
Concentration of HCO3- at 30 minutes after recanalization | 30 minutes after recanalization
Concentration of base excess at 30 minutes after recanalization | 30 minutes after recanalization
partial pressure of oxygen at 30 minutes after recanalization | 30 minutes after recanalization
partial pressure of carbon dioxide at 30 minutes after recanalization | 30 minutes after recanalization
pH value immediately after recanalization | about 1 minute after recanalization
Concentration of HCO3- immediately after recanalization | about 1 minute after recanalization
Concentration of base excess immediately after recanalization | about 1 minute after recanalization
partial pressure of oxygen immediately after recanalization | about 1 minute after recanalization
partial pressure of carbon dioxide immediately after recanalization | about 1 minute after recanalization
Concentration of serum interleukin-6 at 30 minutes after recanalization | 30 minutes after recanalization
Concentration of serum tumor necrosis factor α at 30 minutes after recanalization | 30 minutes after recanalization
Concentration of serum brain-derived neurotrophic factor at 30 minutes after recanalization | 30 minutes after recanalization
score of modified Rankin's scale at 24 hours after recanalization | 24 hours after recanalization
  the minimum and maximum values of modified Rankin's scale is 0 and 5, and higher scores mean a worse outcome.
incidence of stroke during hospitalization | From end of surgery to discharge from hospital, at an average of 5 days
Incidence of death during hospitalization | From end of surgery to discharge from hospital, at an average of 5 days
length of hospitalization | From end of surgery to discharge from hospital, at an average of 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of the Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garzelli L, Nuzzo A, Hamon A, Ben Abdallah I, Gregory J, Raynaud L, Paulatto L, Dioguardi Burgio M, Castier Y, Panis Y, Vilgrain V, Corcos O, Ronot M. Reperfusion injury on computed tomography following endovascular revascularization of acute mesenteric ischemia: prevalence, risk factors, and patient outcome. Insights Imaging. 2022 Dec 13;13(1):194. doi: 10.1186/s13244-022-01339-9. PMID 36512135
- [Result] Onalan A, Gurkas E, Akpinar CK, Dogan H, Acar T, Acar B, Aykac O, Uysal Kocabas Z, Balgetir F, Ozdemir AO. Arterial blood gas analysis predicts futile recanalization in mechanical thrombectomy-treated acute ischemic stroke patients: a multicenter study. Eur Rev Med Pharmacol Sci. 2024 Feb;28(4):1594-1604. doi: 10.26355/eurrev_202402_35488. PMID 38436197